CLINICAL TRIAL: NCT03862638
Title: Yoga Therapy for Chronic Tension-Type Headache: An Evaluation Study
Brief Title: Yoga Therapy for Chronic Tension-Type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Yog-Kulam (Other); Department of Zoology, University of Rajasthan, India (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMP/23891
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Chronic Tension-Type Headache
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Therapy (Experimental): Yoga therapy session lasted for 60 minutes consisting physical posture, Breath work, Relaxation, guided meditation, chants and combination techniques for groups sessions.
  Interventions: Other: Yoga Therapy

INTERVENTIONS:
Other: Yoga Therapy — Yoga therapy is therapeutic application of yoga, specifically designed to treat the condition using physical posture, breathing exercises, guided relaxation and meditation.
  Other Names: Yoga

SUMMARY:
Chronic tension headache represents a considerable social burden in terms of both costs to the health services and also the costs of lost productivity. Episodic tension-type headache can be treated with rest and analgesics, while chronic tension-type headache demands a more fundamental treatment.

Effectiveness of yoga therapy in the management of chronic tension type headache is limited. In this study, yoga therapy was used to explore its effect on chronic tension-type headache.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria of CTTH in the international classification of headache disorders, 3rd edition (beta version) (ICHD-III beta);
* Aged 18-55 years;
* Having the ability of understanding and completing the headache dairy;
* Provide written informed consent.

Exclusion Criteria:

* No headache during the pervious 3 months;
* Taking any prophylactic medication during the previous one month;
* Secondary headache or any systematic cause
* Having serious conditions of the heart, liver, kidney or other organs;
* In pregnancy or lactation, or planning to be pregnant in 6 months;
* Drug and Substance abuse
* Diagnosed psychiatric condition
* Taking any other complementary and alternative medicines
* Practicing yoga of any kind in last three months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2010-04-10 (Actual); Primary Completion 2012-12-12 (Actual); Study Completion 2013-01-15 (Actual)

PRIMARY OUTCOMES:
The number of days with headache | Change from baseline to 12-week of intervention
  Number of days with headache every four weeks were assessed through headache diaries

SECONDARY OUTCOMES:
The medication intake | Change from baseline to 12 week of intervention
  Medication score per month were recorded through headache diaries
Intensity of Pan | Change from baseline to12 week of intervention
  Each headache intensity was measure through 0-10 scale; 0 was no pain and 10 was worst pain
Duration of Pain | Change from baseline to12 week of intervention
  Duration of each headache was measured through headache diaries

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Yog-Kulam; PJ John, PhD, Study Director — Deaprtment of Zoology, University of Rajasthan; Chandra M Sharma, DM, Study Chair — SMS Medical College and Hospital
Locations (1):
- NMP Medical Research Institue, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided